CLINICAL TRIAL: NCT00547248
Title: Booster Vaccination Course With the Pneumococcal Vaccine GSK 1024850A, DTPw-HBV/Hib and OPV or IPV in Children Who Completed the Primary Vaccination Course in Study 107007
Brief Title: Pneumococcal Vaccine Booster Study in Healthy Children 12-18 Mths Old Previously Primed With the Same Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109509
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Booster vaccination.; Immunogenicity; Pneumococcal vaccine; Safety; Pneumococcal disease
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; Tritanrix-HepB vaccine; Hiberix; HibTITER protein, Haemophilus influenzae; Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (4):
- Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group (Experimental): Subjects in the Philippines, primary vaccinated at 6-10-14 weeks of age, receiving booster dose of Synflorix™ vaccine, co-administered with Tritanrix™-HepB/ Hiberix™ and Polio Sabin™ vaccines at 12-18 months of age.
  Interventions: Biological: Synflorix; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin
- Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group (Active Comparator): Subjects in the Philippines, primary vaccinated at 6-10-14 weeks of age, receiving booster dose of the Prevenar™ vaccine, co-administered with Tritanrix™-HepB/ Hiberix™ and Polio Sabin™ at 12-18 months of age.
  Interventions: Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Polio Sabin; Biological: Prevenar (Wyeth)
- Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group (Experimental): Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of Synflorix™ vaccine co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ vaccines at 12-18 months of age.
  Interventions: Biological: Synflorix; Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Poliorix
- Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group (Active Comparator): Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of the Prevenar™ vaccine, co-administered with Tritanrix -HepB/ Hiberix and Poliorix™ at 12-18 months of age.
  Interventions: Biological: Tritanrix-HepB; Biological: Hiberix; Biological: Poliorix; Biological: Prevenar (Wyeth)

INTERVENTIONS:
Biological: Synflorix — Intramuscular injection, 1 dose
  Other Names: Pneumococcal conjugate vaccine GSK1024850A
  Arms: Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group; Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group
Biological: Tritanrix-HepB — Intramuscular injection, 1 dose
  Other Names: DTPw-HBV vaccine
Biological: Hiberix — Reconstituted with Tritanrix-Hep B before injection
  Other Names: Hib vaccine
Biological: Polio Sabin — Oral, 1 dose
  Other Names: OPV
  Arms: Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group; Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group
Biological: Poliorix — Intramuscular injection, 1 dose
  Other Names: IPV
  Arms: Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group; Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group
Biological: Prevenar (Wyeth) — Intramuscular injection, 1 dose
  Other Names: Pneumococcal conjugate vaccine
  Arms: Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group; Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group

SUMMARY:
The purpose of this observer blind study is to assess the safety in terms of fever >39°C (rectal temperature) and the immunogenicity in terms of antibody response following a booster vaccination with pneumococcal vaccine GSK 1024850A at 12 to 18 months of age in children previously primed with the same vaccines including a pneumococcal conjugate vaccine co-administered with a diphtheria, tetanus, whole cell pertussis (DTPw)-combined vaccine and OPV or IPV vaccines. Subjects participating in this study should have received three doses of pneumococcal conjugate vaccine in the primary study.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00344318)

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 12-18 months of age at the time of the booster vaccination and who previously participated in study 107007 and received three doses of pneumococcal conjugate vaccine.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period (active phase and extended safety follow-up), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within one month preceding the booster dose of study vaccines, or planned use during the entire study period
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the booster dose of study vaccines.
* Planned administration/administration of a vaccine not foreseen by the study protocol, during the period starting one month before the booster dose of study vaccines and up to the follow-up visit.
* Administration of any pneumococcal, diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b vaccine other than the study vaccines from study 107007.
* History of, or intercurrent diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b diseases.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or progressive neurological disease.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products within three months preceding the booster dose of study vaccines or planned administration during the active phase of the study.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 756 (Actual)
Dates: Start 2007-10-22 (Actual); Primary Completion 2008-05-10 (Actual); Study Completion 2008-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, City of Muntinlupa, Philippines
- Poland (5):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Tuchola
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bermal N, Szenborn L, Edison A, Hernandez M, Pejcz J, Majda-Stanislawska E, Gatchalian S, Fanic A, Dieussaert I, Schuerman L. Safety and immunogenicity of a booster dose of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine coadministered with DTPw-HBV/Hib and poliovirus vaccines. Pediatr Infect Dis J. 2011 Jan;30(1):69-72. doi: 10.1097/INF.0b013e3181f2da06. PMID 20980933
- [Background] Bermal N et al. Primary and booster vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine (PHiD-CV) co-administered with DTPw-HBV/Hib and polio vaccines. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Nancy B et al. Booster dose of 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) administered to children in the Philippines: antibody responses and safety. Abstract presented at the 13th Asian Pacific Congress of Pediatrics (APCP). Shanghai, China, 14-18 October 2009.
- [Background] Schuerman L et al. Immune responses against cross-reactive pneumococcal serotypes 6A and 19A with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Immune responses to the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) appear not influenced by co-administration with DTPw-combination vaccine. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group: Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of the Prevenar™ vaccine, co-administered with Tritanrix -HepB/ Hiberix and Poliorix at 12-18 months of age.
Period: Overall Study
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Started | 280 | 93 | 285 | 98
Completed | 280 | 93 | 275 | 96
Not Completed | 0 | 0 | 10 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Migrated/moved from study area | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Prevenar + Tritanrix - HepB/ Hiberix + Poliorix Group: Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of the Prevenar™ vaccine, co-administered with Tritanrix -HepB/ Hiberix™ and Poliorix™ at 12-18 months of age.
- Total: Total of all reporting groups
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix - HepB/ Hiberix + Poliorix Group | Total
Number analyzed (Participants) | 280 | 93 | 285 | 98 | 756
Age, Continuous [Geometric Mean (Standard Deviation); unit: Months] | 16.2 (0.66) | 16.2 (0.59) | 17.2 (0.84) | 17.2 (0.88) | 16.71 (0.90)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Categorical: Female | 133 | 43 | 134 | 43 | 353
  Gender Categorical: Male | 147 | 50 | 151 | 55 | 403
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: White - Caucasian / European heritage | 0 | 0 | 285 | 98 | 383
  Geographic ancestry: Asian - south east Asian heritage | 280 | 93 | 0 | 0 | 373

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Rectal Temperature Greater Than (>) the Cut-off
Description: Fever was measured as rectal temperature. The cut-off was 39.0 degree Celsius (°C). Assessment of occurrences of fever > 39.0 (°C) was performed after booster vaccination with Synflorix™ or Prevenar™ vaccines.
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with the symptom sheets filled in. For the purpose of the analysis, subjects were pooled into two groups, according to the booster vaccine they have received (Synflorix™ or Prevenar™).
Measure: Count of Participants; unit: Participants
Groups:
- Synflorix Pooled Group: Subjects primary vaccinated at 6-10-14 weeks of age, receiving a booster dose of Synflorix™ vaccine, either co-administered with Tritanrix™-HepB/ Hiberix™ and Polio Sabin™ vaccines in the Philippines or co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ vaccines in Poland, at 12-18 months of age.
- Prevenar Pooled Group: Subjects primary vaccinated at 6-10-14 weeks of age, receiving a booster dose of the Prevenar™ vaccine, either co-administered with Tritanrix™-HepB/ Hiberix™ and Polio Sabin™ vaccines in the Philippines or co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ vaccines in Poland, at 12-18 months of age.
Arm/Group | Synflorix Pooled Group | Prevenar Pooled Group
Number analyzed (Participants) | 558 | 189
Participants | 64 | 20
Statistical Analysis 1: Comparison: Synflorix Pooled Group vs Prevenar Pooled Group; Test type: Non-Inferiority — Non-inferiority was demonstrated if the difference in terms of incidence of post-immunization febrile reactions (rectal temperature > 39.0°C) in Synflorix™ vaccine minus Prevenar™ did not exceed the pre-defined clinically acceptable threshold of 5% + half the incidence in Prevenar; Philips' statistical test; Difference in percentage = 0.89, 95% CI 2-sided [-4.82 to 5.59]

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. "Any" was defined as incidence of the specified symptom regardless of intensity. Grade 3 pain was defined as crying when limb was moved/ spontaneously painful. Grade 3 swelling/ redness was defined as swelling/ redness greater than (>) 30 millimeters (mm).
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Groups:
- Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group: Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of the Prevenar™ vaccine, co-administered with Tritanrix -HepB/ Hiberix™ and Poliorix™ at 12-18 months of age.
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 280 | 93 | 278 | 96
Participants
  Any Pain | 203 | 66 | 248 | 77
  Grade 3 Pain | 40 | 20 | 117 | 39
  Any Redness | 107 | 37 | 197 | 66
  Grade 3 Redness | 8 | 3 | 35 | 11
  Any Swelling | 92 | 32 | 158 | 52
  Grade 3 Swelling | 21 | 9 | 34 | 8

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature greater than or equal to (≥) 38.0°C), irritability, and loss of appetite."Any" was defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) >40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/ preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all.
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 280 | 93 | 278 | 96
Participants
  Any Drowsiness | 90 | 32 | 190 | 66
  Grade 3 Drowsiness | 5 | 1 | 7 | 2
  Any Fever | 138 | 51 | 215 | 65
  Grade 3 Fever | 0 | 0 | 1 | 0
  Any Irritability | 173 | 64 | 243 | 79
  Grade 3 Irritability | 12 | 3 | 40 | 5
  Any Loss of appetite | 97 | 28 | 184 | 57
  Grade 3 Loss of appetite | 8 | 1 | 13 | 1

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 280 | 93 | 285 | 98
Participants | 25 | 9 | 106 | 35

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: Throughout the active phase of the study (Month 0 to Month 1)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 280 | 93 | 285 | 98
Participants | 2 | 0 | 5 | 2

6. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off
Description: The cut-off was 0.20 microgram per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence, which included all subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sampling taken before the administration of the study booster dose (pre-booster blood sampling).
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 130 | 44
Participants
  Anti-1, Month 0: number analyzed (Participants) | 136 | 42 | 128 | 40
  Anti-1, Month 0 | 100 | 2 | 64 | 2
  Anti-1, Month 1: number analyzed (Participants) | 136 | 42 | 128 | 40
  Anti-1, Month 1 | 136 | 3 | 125 | 2
  Anti-4, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-4, Month 0 | 113 | 25 | 78 | 23
  Anti-4, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-4, Month 1 | 136 | 43 | 125 | 43
  Anti-5, Month 0: number analyzed (Participants) | 135 | 42 | 129 | 42
  Anti-5, Month 0 | 118 | 7 | 98 | 3
  Anti-5, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-5, Month 1 | 136 | 8 | 124 | 3
  Anti-6B, Month 0: number analyzed (Participants) | 135 | 43 | 129 | 44
  Anti-6B, Month 0 | 113 | 24 | 90 | 27
  Anti-6B, Month 1: number analyzed (Participants) | 136 | 42 | 125 | 43
  Anti-6B, Month 1 | 134 | 42 | 122 | 41
  Anti-7F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-7F, Month 0 | 128 | 7 | 118 | 1
  Anti-7F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-7F, Month 1 | 136 | 9 | 125 | 1
  Anti-9V, Month 0: number analyzed (Participants) | 135 | 42 | 130 | 44
  Anti-9V, Month 0 | 132 | 40 | 116 | 42
  Anti-9V, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-9V, Month 1 | 136 | 43 | 125 | 43
  Anti-14, Month 0: number analyzed (Participants) | 134 | 43 | 130 | 43
  Anti-14, Month 0 | 126 | 42 | 111 | 40
  Anti-14, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-14, Month 1 | 135 | 43 | 125 | 43
  Anti-18C, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-18C, Month 0 | 130 | 36 | 111 | 35
  Anti-18C, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-18C, Month 1 | 136 | 43 | 125 | 43
  Anti-19F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-19F, Month 0 | 129 | 11 | 121 | 22
  Anti-19F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-19F, Month 1 | 136 | 43 | 123 | 43
  Anti-23F, Month 0: number analyzed (Participants) | 133 | 43 | 130 | 44
  Anti-23F, Month 0 | 123 | 32 | 89 | 40
  Anti-23F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-23F, Month 1 | 135 | 42 | 123 | 42

7. Secondary Outcome: Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations
Description: Seropositivity status, defined as anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence, which included all subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sampling taken before the administration of the study booster dose (pre-booster blood sampling.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 130 | 44
μg/mL
  Anti-1, Month 0: number analyzed (Participants) | 136 | 42 | 128 | 40
  Anti-1, Month 0 | 0.35 [0.29 to 0.42] | 0.03 [0.03 to 0.04] | 0.19 [0.16 to 0.22] | 0.04 [0.03 to 0.05]
  Anti-1, Month 1: number analyzed (Participants) | 136 | 42 | 125 | 43
  Anti-1, Month 1 | 10.8 [9.22 to 12.66] | 0.04 [0.03 to 0.05] | 2.14 [1.8 to 2.55] | 0.04 [0.03 to 0.05]
  Anti-4, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-4, Month 0 | 0.55 [0.45 to 0.67] | 0.34 [0.25 to 0.45] | 0.27 [0.22 to 0.33] | 0.24 [0.19 to 0.3]
  Anti-4, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-4, Month 1 | 13.16 [11.43 to 15.14] | 11.84 [8.74 to 16.04] | 4.21 [3.61 to 4.91] | 6.86 [5.39 to 8.73]
  Anti-5, Month 0: number analyzed (Participants) | 135 | 42 | 129 | 42
  Anti-5, Month 0 | 0.55 [0.47 to 0.64] | 0.06 [0.04 to 0.09] | 0.4 [0.34 to 0.47] | 0.04 [0.03 to 0.05]
  Anti-5, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-5, Month 1 | 14.59 [12.53 to 16.99] | 0.09 [0.06 to 0.13] | 2.54 [2.11 to 3.06] | 0.05 [0.04 to 0.06]
  Anti-6B, Month 0: number analyzed (Participants) | 135 | 43 | 129 | 44
  Anti-6B, Month 0 | 0.66 [0.54 to 0.8] | 0.38 [0.22 to 0.65] | 0.34 [0.28 to 0.41] | 0.34 [0.2 to 0.59]
  Anti-6B, Month 1: number analyzed (Participants) | 136 | 42 | 125 | 43
  Anti-6B, Month 1 | 7.02 [5.83 to 8.45] | 9.08 [6.5 to 12.7] | 2.31 [1.93 to 2.75] | 6.28 [4.18 to 9.44]
  Anti-7F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-7F, Month 0 | 0.9 [0.77 to 1.04] | 0.05 [0.03 to 0.07] | 0.58 [0.51 to 0.67] | 0.03 [0.03 to 0.04]
  Anti-7F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-7F, Month 1 | 12.52 [11.09 to 14.13] | 0.06 [0.04 to 0.1] | 4.14 [3.61 to 4.74] | 0.03 [0.03 to 0.04]
  Anti-9V, Month 0: number analyzed (Participants) | 135 | 42 | 130 | 44
  Anti-9V, Month 0 | 1.16 [0.98 to 1.37] | 0.77 [0.59 to 0.99] | 0.59 [0.5 to 0.7] | 0.58 [0.47 to 0.71]
  Anti-9V, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-9V, Month 1 | 14.42 [12.44 to 16.7] | 20.31 [15.44 to 26.71] | 4.63 [4 to 5.36] | 13.6 [11.12 to 16.62]
  Anti-14, Month 0: number analyzed (Participants) | 134 | 43 | 130 | 43
  Anti-14, Month 0 | 1.32 [1.07 to 1.63] | 1.83 [1.26 to 2.66] | 0.84 [0.66 to 1.07] | 1.04 [0.75 to 1.43]
  Anti-14, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-14, Month 1 | 17.07 [14.12 to 20.64] | 27.42 [20.96 to 35.86] | 5.93 [4.97 to 7.09] | 15.51 [12.14 to 19.82]
  Anti-18C, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-18C, Month 0 | 1.43 [1.2 to 1.71] | 0.42 [0.32 to 0.55] | 0.63 [0.52 to 0.77] | 0.4 [0.3 to 053]
  Anti-18C, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-18C, Month 1 | 39.59 [34.04 to 46.05] | 12.07 [9.23 to 15.79] | 10.49 [8.81 to 12.49] | 9.92 [7.74 to 12.71]
  Anti-19F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-19F, Month 0 | 1.33 [1.08 to 1.64] | 0.16 [0.1 to 0.26] | 0.99 [0.81 to 1.22] | 0.35 [0.2 to 0.61]
  Anti-19F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-19F, Month 1 | 21.25 [18.07 to 24.98] | 6.61 [4.9 to 8.92] | 12.23 [9.89 to 15.13] | 6.01 [4.75 to 7.6]
  Anti-23F, Month 0: number analyzed (Participants) | 133 | 43 | 130 | 44
  Anti-23F, Month 0 | 0.94 [0.76 to 1.16] | 0.41 [0.26 to 0.64] | 0.33 [0.27 to 0.4] | 0.62 [0.43 to 0.91]
  Anti-23F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-23F, Month 1 | 13.47 [11.38 to 15.94] | 14.78 [9.45 to 23.11] | 3.16 [2.61 to 3.83] | 10.77 [7.19 to 16.12]

8. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 125 | 37
Titers
  OPA Anti-1, Month 0: number analyzed (Participants) | 134 | 43 | 122 | 37
  OPA Anti-1, Month 0 | 13.2 [10.2 to 16.9] | 4.6 [3.9 to 5.4] | 8.5 [7 to 10.5] | 4.7 [3.8 to 5.8]
  OPA Anti-1, Month 1: number analyzed (Participants) | 134 | 43 | 120 | 37
  OPA Anti-1, Month 1 | 1571.6 [1210.7 to 2040] | 4.9 [4.1 to 5.8] | 161.4 [120.7 to 215.9] | 5.4 [4 to 7.4]
  OPA Anti-4, Month 0: number analyzed (Participants) | 127 | 42 | 114 | 33
  OPA Anti-4, Month 0 | 40.5 [27.6 to 59.2] | 18.5 [10 to 34.2] | 12.5 [8.9 to 17.4] | 12.4 [6.7 to 22.8]
  OPA Anti-4, Month 1: number analyzed (Participants) | 134 | 43 | 119 | 35
  OPA Anti-4, Month 1 | 5035.8 [4214 to 6017.8] | 4783.5 [3432 to 6667.2] | 2498.7 [2103.3 to 2968.4] | 4812.5 [3167.8 to 7311.3]
  OPA Anti-5, Month 0: number analyzed (Participants) | 133 | 43 | 119 | 36
  OPA Anti-5, Month 0 | 19.8 [16 to 24.7] | 4.2 [3.8 to 4.6] | 10.9 [8.8 to 13.6] | 4.5 [3.7 to 5.5]
  OPA Anti-5, Month 1: number analyzed (Participants) | 130 | 43 | 117 | 36
  OPA Anti-5, Month 1 | 1135.8 [928.5 to 1389.6] | 4.9 [3.9 to 6] | 149.1 [115.4 to 192.5] | 4.3 [3.8 to 4.8]
  OPA Anti-6B, Month 0: number analyzed (Participants) | 132 | 43 | 124 | 37
  OPA Anti-6B, Month 0 | 97.8 [61.5 to 155.5] | 56.6 [21.3 to 150.1] | 9.9 [7.2 to 13.5] | 23.3 [9.1 to 60.1]
  OPA Anti-6B, Month 1: number analyzed (Participants) | 136 | 43 | 120 | 35
  OPA Anti-6B, Month 1 | 2896.8 [2247.5 to 3733.8] | 9302.7 [7187.3 to 12040.8] | 405.3 [267.4 to 614.3] | 3547.1 [1500.7 to 8384.5]
  OPA Anti-7F, Month 0: number analyzed (Participants) | 135 | 41 | 116 | 31
  OPA Anti-7F, Month 0 | 2278.4 [1803.1 to 2879] | 378.8 [136.9 to 1048] | 796.3 [582.2 to 1089.1] | 63.6 [21.3 to 190.1]
  OPA Anti-7F, Month 1: number analyzed (Participants) | 136 | 42 | 122 | 24
  OPA Anti-7F, Month 1 | 12484 [10750.7 to 14496.8] | 1407.7 [694.6 to 2852.9] | 6436.1 [5507.6 to 7521] | 90.6 [25.2 to 325.5]
  OPA Anti-9V, Month 0: number analyzed (Participants) | 136 | 42 | 122 | 37
  OPA Anti-9V, Month 0 | 788 [655.1 to 947.8] | 666.8 [482.1 to 922.2] | 380.2 [313.1 to 461.7] | 247.5 [164.9 to 371.3]
  OPA Anti-9V, Month 1: number analyzed (Participants) | 134 | 42 | 121 | 35
  OPA Anti-9V, Month 1 | 4842 [4122.7 to 5686.9] | 7387.8 [5429.2 to 10052.9] | 3499.9 [2950.8 to 4151.3] | 6881.4 [4883.6 to 9696.4]
  OPA Anti-14, Month 0: number analyzed (Participants) | 130 | 42 | 106 | 31
  OPA Anti-14, Month 0 | 298.4 [220.1 to 404.7] | 337.2 [207 to 549.2] | 179.6 [127.4 to 253.2] | 236.6 [132.6 to 422.2]
  OPA Anti-14, Month 1: number analyzed (Participants) | 132 | 42 | 120 | 36
  OPA Anti-14, Month 1 | 3579.7 [2966.3 to 4319.9] | 4097.3 [3019.2 to 5560.2] | 1961.3 [1630 to 2359.8] | 2939.5 [2022.3 to 4272.7]
  OPA Anti-18C, Month 0: number analyzed (Participants) | 129 | 42 | 121 | 37
  OPA Anti-18C, Month 0 | 19.8 [15.2 to 25.9] | 4.5 [3.9 to 5.2] | 7.8 [6.5 to 9.4] | 4.5 [4 to 5.2]
  OPA Anti-18C, Month 1: number analyzed (Participants) | 134 | 43 | 115 | 36
  OPA Anti-18C, Month 1 | 2417.2 [1989.9 to 2936.2] | 966.5 [607.1 to 1538.6] | 694 [532.9 to 903.7] | 612.1 [338.4 to 1107]
  OPA Anti-19F, Month 0: number analyzed (Participants) | 135 | 43 | 125 | 37
  OPA Anti-19F, Month 0 | 58.6 [45.2 to 76] | 7.3 [4.5 to 11.8] | 33.3 [25.7 to 43.2] | 11.1 [6 to 20.6]
  OPA Anti-19F, Month 1: number analyzed (Participants) | 136 | 42 | 122 | 37
  OPA Anti-19F, Month 1 | 2016 [1609 to 2526] | 473.2 [263.5 to 849.9] | 1059.8 [808.2 to 1389.7] | 471 [270 to 821.8]
  OPA Anti-23F, Month 0: number analyzed (Participants) | 136 | 43 | 118 | 36
  OPA Anti-23F, Month 0 | 948.9 [688.4 to 1308.2] | 661.9 [312.5 to 1402] | 301.8 [198.4 to 459] | 790.6 [326.8 to 1912.6]
  OPA Anti-23F, Month 1: number analyzed (Participants) | 136 | 43 | 121 | 37
  OPA Anti-23F, Month 1 | 7456.2 [6301.9 to 8822] | 23177.9 [13235.9 to 40587.7] | 3427.3 [2727.7 to 4306.3] | 19943.3 [13473.1 to 29520.5]

9. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD)
Description: Seropositivity status, defined as anti-PD antibody concentrations ≥100 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 135 | 43 | 128 | 43
EL.U/mL
  Anti-PD, Month 0: number analyzed (Participants) | 132 | 43 | 128 | 43
  Anti-PD, Month 0 | 573.1 [495.7 to 662.6] | 136.8 [102 to 183.3] | 526.8 [427.4 to 649.3] | 73.8 [58.4 to 93.2]
  Anti-PD, Month 1: number analyzed (Participants) | 135 | 43 | 125 | 43
  Anti-PD, Month 1 | 4973.9 [4280.2 to 5780] | 124.1 [92.8 to 166] | 2769.6 [2308.5 to 3322.7] | 91.6 [72 to 116.7]

10. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: Seropositivity status, defined as anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 130 | 44
μg/mL
  Anti-6A, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 43
  Anti-6A, Month 0 | 0.46 [0.36 to 0.6] | 0.24 [0.14 to 0.4] | 0.12 [0.1 to 0.14] | 0.13 [0.08 to 0.2]
  Anti-6A, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-6A, Month 1 | 4.07 [3.09 to 5.36] | 4.57 [2.92 to 7.17] | 0.84 [0.65 to 1.08] | 2.54 [1.65 to 3.93]
  Anti-19A, Month 0: number analyzed (Participants) | 134 | 43 | 130 | 44
  Anti-19A, Month 0 | 0.24 [0.19 to 0.3] | 0.08 [0.05 to 0.12] | 0.16 [0.12 to 0.2] | 0.06 [0.04 to 0.08]
  Anti-19A, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-19A, Month 1 | 3.22 [2.46 to 4.21] | 0.58 [0.37 to 0.91] | 1.75 [1.27 to 2.43] | 0.38 [0.25 to 0.58]

11. Secondary Outcome: Opsonophagocytic Activity (OPA) Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A ≥ 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 134 | 43 | 123 | 36
Titers
  OPA Anti-6A, Month 0: number analyzed (Participants) | 117 | 39 | 108 | 32
  OPA Anti-6A, Month 0 | 113.6 [73.6 to 175.4] | 191.4 [89.7 to 408.2] | 46.8 [30.8 to 71.1] | 42.2 [19.3 to 92.1]
  OPA Anti-6A, Month 1: number analyzed (Participants) | 133 | 43 | 109 | 32
  OPA Anti-6A, Month 1 | 882.8 [665.9 to 1170.3] | 2563.8 [1689.9 to 3889.4] | 369.7 [258.5 to 528.8] | 1394.5 [827.9 to 2348.9]
  OPA Anti-19A, Month 0 | 5.3 [4.5 to 6.3] | 5.1 [3.6 to 7.3] | 5.3 [4.5 to 6.2] | 4.4 [3.6 to 5.3]
  OPA Anti-19A, Month 1: number analyzed (Participants) | 133 | 40 | 115 | 32
  OPA Anti-19A, Month 1 | 89.3 [58.9 to 135.4] | 8.7 [5.4 to 14.2] | 70.7 [45.3 to 110.4] | 20.3 [8.8 to 46.8]

12. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F Antibody Concentrations ≥ the Cut-off
Description: The cut-off of the assay was 0.05 μg/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 130 | 44
Participants
  Anti-1, Month 0: number analyzed (Participants) | 136 | 42 | 128 | 40
  Anti-1, Month 0 | 135 | 7 | 122 | 8
  Anti-1, Month 1: number analyzed (Participants) | 136 | 42 | 125 | 43
  Anti-1, Month 1 | 136 | 11 | 125 | 9
  Anti-4, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-4, Month 0 | 134 | 43 | 126 | 42
  Anti-4, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-4, Month 1 | 136 | 43 | 125 | 43
  Anti-5, Month 0: number analyzed (Participants) | 135 | 42 | 129 | 42
  Anti-5, Month 0 | 135 | 18 | 128 | 13
  Anti-5, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-5, Month 1 | 136 | 31 | 125 | 20
  Anti-6B, Month 0: number analyzed (Participants) | 135 | 43 | 129 | 44
  Anti-6B, Month 0 | 132 | 40 | 127 | 39
  Anti-6B, Month 1: number analyzed (Participants) | 136 | 42 | 125 | 43
  Anti-6B, Month 1 | 135 | 42 | 124 | 42
  Anti-7F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 42
  Anti-7F, Month 0 | 135 | 13 | 130 | 8
  Anti-7F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-7F, Month 1 | 136 | 17 | 125 | 11
  Anti-9V, Month 0: number analyzed (Participants) | 135 | 42 | 130 | 44
  Anti-9V, Month 0 | 135 | 42 | 130 | 44
  Anti-9V, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-9V, Month 1 | 136 | 43 | 125 | 43
  Anti-14, Month 0: number analyzed (Participants) | 134 | 43 | 130 | 43
  Anti-14, Month 0 | 134 | 42 | 130 | 43
  Anti-14, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-14, Month 1 | 136 | 43 | 125 | 43
  Anti-18C, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-18C, Month 0 | 135 | 43 | 129 | 44
  Anti-18C, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-18C, Month 1 | 136 | 43 | 125 | 43
  Anti-19F, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 44
  Anti-19F, Month 0 | 134 | 37 | 129 | 43
  Anti-19F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-19F, Month 1 | 136 | 43 | 124 | 43
  Anti-23F, Month 0: number analyzed (Participants) | 133 | 43 | 130 | 44
  Anti-23F, Month 0 | 132 | 40 | 125 | 43
  Anti-23F, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-23F, Month 1 | 136 | 42 | 124 | 42

13. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F ≥ the Cut-off
Description: The cut-off for the assay was 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 125 | 37
Participants
  OPA Anti-1, Month 0: number analyzed (Participants) | 134 | 43 | 122 | 37
  OPA Anti-1, Month 0 | 61 | 3 | 45 | 3
  OPA Anti-1, Month 1: number analyzed (Participants) | 134 | 43 | 120 | 37
  OPA Anti-1, Month 1 | 134 | 5 | 114 | 5
  OPA Anti-4, Month 0: number analyzed (Participants) | 127 | 42 | 114 | 33
  OPA Anti-4, Month 0 | 83 | 20 | 39 | 12
  OPA Anti-4, Month 1: number analyzed (Participants) | 134 | 43 | 119 | 35
  OPA Anti-4, Month 1 | 134 | 43 | 119 | 35
  OPA Anti-5, Month 0: number analyzed (Participants) | 133 | 43 | 119 | 36
  OPA Anti-5, Month 0 | 94 | 1 | 56 | 2
  OPA Anti-5, Month 1: number analyzed (Participants) | 130 | 43 | 117 | 36
  OPA Anti-5, Month 1 | 130 | 4 | 114 | 1
  OPA Anti-6B, Month 0: number analyzed (Participants) | 132 | 43 | 124 | 37
  OPA Anti-6B, Month 0 | 93 | 21 | 34 | 14
  OPA Anti-6B, Month 1: number analyzed (Participants) | 136 | 43 | 120 | 35
  OPA Anti-6B, Month 1 | 134 | 43 | 106 | 32
  OPA Anti-7F, Month 0: number analyzed (Participants) | 135 | 41 | 116 | 31
  OPA Anti-7F, Month 0 | 133 | 28 | 109 | 15
  OPA Anti-7F, Month 1: number analyzed (Participants) | 136 | 40 | 122 | 24
  OPA Anti-7F, Month 1 | 136 | 36 | 122 | 13
  OPA Anti-9V, Month 0: number analyzed (Participants) | 136 | 42 | 122 | 37
  OPA Anti-9V, Month 0 | 135 | 42 | 121 | 36
  OPA Anti-9V, Month 1: number analyzed (Participants) | 134 | 42 | 121 | 35
  OPA Anti-9V, Month 1 | 134 | 42 | 121 | 35
  OPA Anti-14, Month 0: number analyzed (Participants) | 130 | 42 | 106 | 31
  OPA Anti-14, Month 0 | 119 | 39 | 93 | 29
  OPA Anti-14, Month 1: number analyzed (Participants) | 132 | 42 | 120 | 36
  OPA Anti-14, Month 1 | 132 | 42 | 120 | 36
  OPA Anti-18C, Month 0: number analyzed (Participants) | 129 | 42 | 121 | 37
  OPA Anti-18C, Month 0 | 84 | 3 | 42 | 4
  OPA Anti-18C, Month 1: number analyzed (Participants) | 134 | 43 | 115 | 36
  OPA Anti-18C, Month 1 | 133 | 42 | 114 | 36
  OPA Anti-19F, Month 0: number analyzed (Participants) | 135 | 43 | 125 | 37
  OPA Anti-19F, Month 0 | 117 | 7 | 96 | 12
  OPA Anti-19F, Month 1: number analyzed (Participants) | 136 | 42 | 122 | 37
  OPA Anti-19F, Month 1 | 135 | 39 | 118 | 36
  OPA Anti-23F, Month 0: number analyzed (Participants) | 136 | 43 | 118 | 36
  OPA Anti-23F, Month 0 | 130 | 37 | 99 | 30
  OPA Anti-23F, Month 1: number analyzed (Participants) | 136 | 43 | 121 | 37
  OPA Anti-23F, Month 1 | 136 | 42 | 120 | 37

14. Secondary Outcome: Number of Subjects With Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A ≥ the Cut-off
Description: The cut-of for the assay was 0.05 μg/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 136 | 43 | 130 | 44
Participants
  Anti-6A, Month 0: number analyzed (Participants) | 135 | 43 | 130 | 43
  Anti-6A, Month 0 | 128 | 37 | 105 | 33
  Anti-6A, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-6A, Month 1 | 133 | 42 | 125 | 42
  Anti-19A, Month 0: number analyzed (Participants) | 134 | 43 | 130 | 44
  Anti-19A, Month 0 | 124 | 25 | 105 | 27
  Anti-19A, Month 1: number analyzed (Participants) | 136 | 43 | 125 | 43
  Anti-19A, Month 1 | 135 | 42 | 119 | 42

15. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity (OPA) Against Pneumococcal Cross-reactive Serotypes 6A and 19A ≥ the Cut-off
Description: The cut-off for the assay was 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 134 | 43 | 123 | 36
Participants
  OPA Anti-6A, Month 0: number analyzed (Participants) | 117 | 39 | 108 | 32
  OPA Anti-6A, Month 0 | 82 | 30 | 63 | 19
  OPA Anti-6A, Month 1: number analyzed (Participants) | 133 | 43 | 109 | 32
  OPA Anti-6A, Month 1 | 127 | 43 | 97 | 32
  OPA Anti-19A, Month 0 | 14 | 2 | 11 | 1
  OPA Anti-19A, Month 1: number analyzed (Participants) | 133 | 40 | 115 | 32
  OPA Anti-19A, Month 1 | 92 | 11 | 74 | 12

16. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Protein D (Anti-PD) ≥ the Cut-off
Description: The cut-off for the assay was 100 ELISA units per milliliter (EL.U/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 135 | 43 | 128 | 43
Participants
  Anti-PD, Month 0: number analyzed (Participants) | 132 | 43 | 128 | 43
  Anti-PD, Month 0 | 131 | 28 | 117 | 11
  Anti-PD, Month 1: number analyzed (Participants) | 135 | 43 | 125 | 43
  Anti-PD, Month 1 | 135 | 23 | 125 | 19

17. Secondary Outcome: Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Seroprotection status, defined as anti-diphtheria toxoid or anti-tetanus toxoid antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
IU/mL
  Anti-DT, Month 0 | 0.258 [0.209 to 0.319] | 0.17 [0.118 to 0.243] | 0.188 [0.153 to 0.231] | 0.126 [0.088 to 0.179]
  Anti-DT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-DT, Month 1 | 7.829 [6.339 to 9.671] | 4.768 [3.699 to 6.145] | 8.463 [7.11 to 10.074] | 4.876 [3.503 to 6.787]
  Anti-TT, Month 0 | 0.735 [0.629 to 0.858] | 0.455 [0.314 to 0.66] | 0.568 [0.432 to 0.748] | 0.525 [0.29 to 0.951]
  Anti-TT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-TT, Month 1 | 20.979 [18.359 to 23.972] | 9.703 [8.173 to 11.518] | 12.171 [9.772 to 15.16] | 6.719 [4.598 to 9.819]

18. Secondary Outcome: Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentrations
Description: Seroprotection status, defined as anti-PRP antibody concentrations ≥ 0.15 μg/mL and ≥ 1.0 μg/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Synflorix + Tritanrix -HepB/ Hiberix + Poliorix™ Group: Subjects in Poland, primary vaccinated at 2-4-6 months of age, receiving booster dose of Synflorix™ vaccine co-administered with Tritanrix™-HepB/Hiberix™ and Poliorix™ vaccines at 12-18 months of age.
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix™ Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
μg/mL
  Anti-PRP, Month 0 | 5.335 [3.578 to 7.953] | 6.433 [2.93 to 14.124] | 1.03 [0.745 to 1.423] | 0.894 [0.57 to 1.401]
  Anti-PRP, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-PRP, Month 1 | 106.004 [79.937 to 140.572] | 89.376 [55.131 to 144.891] | 53.386 [34.817 to 81.858] | 33.656 [19.464 to 58.198]

19. Secondary Outcome: Anti-Bordetella Pertussis (BPT) Antibody Concentrations
Description: Seropositivity status, defined as anti-BPT antibody concentrations ≥ 15 EL.U/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
EL.U/mL
  Anti-BPT, Month 0 | 12.88 [10.86 to 15.28] | 12.46 [9.32 to 16.65] | 9.54 [8.34 to 10.91] | 10 [8.21 to 12.19]
  Anti-BPT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-BPT, Month 1 | 139.51 [123.26 to 157.89] | 133.45 [110.33 to 161.4] | 121.73 [103.16 to 143.64] | 121.76 [91.81 to 161.47]

20. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations
Description: Seroprotection status, defined as anti-HBs antibody concentrations ≥ 10 milli international units per milliliter (mIU/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 69 | 21 | 64 | 19
mIU/mL
  Anti-HBs, Month 0 | 30 [21.1 to 42.8] | 23.4 [11.5 to 47.7] | 97.9 [77 to 124.5] | 113 [55.1 to 231.7]
  Anti-HBs, Month 1: number analyzed (Participants) | 69 | 21 | 62 | 19
  Anti-HBs, Month 1 | 1220.5 [790.6 to 1884] | 1098.1 [358.4 to 3364.9] | 4428.7 [2980.3 to 6581] | 3188.6 [1171.7 to 8677.1]

21. Secondary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Seroprotection status, defined as anti-polio type 1, anti-polio type 2 and anti-polio type 3 antibody titers ≥ 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix™ Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 69 | 21 | 64 | 20
Titers
  Anti-Polio 1, Month 0: number analyzed (Participants) | 69 | 21 | 63 | 20
  Anti-Polio 1, Month 0 | 329.1 [214.9 to 504.1] | 269 [114.8 to 630.3] | 46.5 [33.6 to 64.4] | 51.1 [28.4 to 91.9]
  Anti-Polio 1, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 1, Month 1 | 854.6 [573.5 to 1273.5] | 426.9 [166.2 to 1096.7] | 932.5 [770.5 to 1128.6] | 727.3 [512.9 to 1059.9]
  Anti-Polio 2, Month 0 | 222.6 [171.8 to 288.3] | 210.4 [115.4 to 383.6] | 50.2 [36.9 to 68.2] | 60.8 [33.4 to 110.8]
  Anti-Polio 2, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 2, Month 1 | 716.9 [487.6 to 1054.1] | 689.1 [304.8 to 1557.9] | 1195.7 [977.8 to 1462.2] | 1206.6 [737 to 1975.4]
  Anti-Polio 3, Month 0 | 102.2 [73.9 to 141.5] | 38.4 [20.3 to 72.9] | 51.8 [37.4 to 71.7] | 71.1 [36.2 to 139.5]
  Anti-Polio 3, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 3, Month 1 | 232.7 [159.6 to 339.4] | 190.4 [78.2 to 463.6] | 1464.2 [1128 to 1900.6] | 1346.2 [857.6 to 2113.2]

22. Secondary Outcome: Number of Subjects With Anti-Bordetella Pertussis (BPT) With Concentrations ≥ the Cut-off
Description: The cut-off for the assay was 15 EL.U/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
Participants
  Anti-BPT, Month 0 | 28 | 10 | 12 | 7
  Anti-BPT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-BPT, Month 1 | 65 | 25 | 59 | 24

23. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations ≥ the Cut-off
Description: The cut-off for the assay was 0.1 milli-international units per milliliter (mIU/mL).
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
Participants
  Anti-DT, Month 0 | 56 | 18 | 49 | 15
  Anti-DT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-DT, Month 1 | 65 | 25 | 59 | 24
  Anti-TT, Month 0 | 65 | 24 | 60 | 23
  Anti-TT, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-TT, Month 1 | 65 | 25 | 58 | 24

24. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration ≥ the Cut-off
Description: The cut-off for the assay was 0.15 μg/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
Participants
  Anti-PRP, Month 0 | 65 | 25 | 58 | 23
  Anti-PRP, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-PRP, Month 1 | 65 | 25 | 59 | 24

25. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentration ≥ the Cut-off
Description: The cut-off for the assay was 1.0 μg/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 65 | 25 | 62 | 24
Participants
  Anti-PRP, Month 0 | 56 | 22 | 32 | 12
  Anti-PRP, Month 1: number analyzed (Participants) | 65 | 25 | 59 | 24
  Anti-PRP, Month 1 | 65 | 25 | 57 | 24

26. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (HBs) Antibody Concentrations ≥ the Cut-off
Description: The cut-off for the assay was 10 mIU/mL.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 69 | 21 | 64 | 19
Participants
  Anti-HBs, Month 0 | 53 | 13 | 63 | 19
  Anti-HBs, Month 1: number analyzed (Participants) | 69 | 21 | 62 | 19
  Anti-HBs, Month 1 | 68 | 19 | 62 | 19

27. Secondary Outcome: Number of Subjects With Anti-polio Type 1, 2 and 3 (Anti-Polio 1, 2 and 3) Antibody Titers ≥ the Cut-off
Description: The cut-off for the assay was 8.
Time Frame: Prior to (Month 0) and one month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 69 | 21 | 64 | 20
Participants
  Anti-Polio 1, Month 0: number analyzed (Participants) | 69 | 21 | 63 | 20
  Anti-Polio 1, Month 0 | 64 | 19 | 56 | 19
  Anti-Polio 1, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 1, Month 1 | 68 | 19 | 63 | 19
  Anti-Polio 2, Month 0 | 69 | 21 | 59 | 19
  Anti-Polio 2, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 2, Month 1 | 69 | 21 | 63 | 19
  Anti-Polio 3, Month 0 | 65 | 17 | 61 | 18
  Anti-Polio 3, Month 1: number analyzed (Participants) | 69 | 21 | 63 | 19
  Anti-Polio 3, Month 1 | 66 | 20 | 63 | 19

28. Secondary Outcome: Number of Subjects With Vaccine Response to Anti-Bordetella Pertussis (BPT)
Description: Vaccine response for anti-BPT, defined as the appearance of antibodies in subjects seronegative at pre-vaccination, or at least 2-fold increase of pre-vaccination antibody concentrations in those who were initially seropositive at pre-vaccination.
Time Frame: One month after booster vaccination (Month 1)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
Number analyzed (Participants) | 37 | 15 | 48 | 16
Participants
  Anti-BPT, S- | 37 | 15 | 48 | 16
  Anti-BPT, S+: number analyzed (Participants) | 28 | 10 | 11 | 7
  Anti-BPT, S+ | 27 | 8 | 11 | 7

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms during the 4-day and unsolicited AEs during the 31- day after booster vaccination; serious adverse events (SAEs): throughout the entire study period from Month 0 to Month 6
Description: The solicited local and general symptoms were only collected for those subjects who filled in their symptom sheets.
Arm/Group | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group
All-Cause Mortality (participants affected / at risk) | 0/280 | 1/93 | 0/285 | 0/98
Serious Adverse Events (participants affected / at risk) | 6/280 | 1/93 | 14/285 | 5/98
Other Adverse Events (participants affected / at risk) | 237/280 | 78/93 | 276/285 | 92/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group (N=280) | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group (N=93) | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group (N=285) | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group (N=98)
Internal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 3 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 5 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 2 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0
Infestation (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix + Tritanrix -HepB/ Hiberix + Polio Sabin Group (N=280) | Prevenar + Tritanrix - HepB/ Hiberix + Polio Sabin Group (N=93) | Synflorix + Tritanrix -HepB/ Hiberix + Poliorix Group (N=285) | Prevenar + Tritanrix -HepB/ Hiberix + Poliorix Group (N=98)
Decreased appetite (Metabolism and nutrition disorders) | 97 (97) | 28 (28) | 184 (184) | 57 (57)
Erythema (Skin and subcutaneous tissue disorders) | 107 (107) | 37 (37) | 197 (197) | 66 (66)
Irritability (Psychiatric disorders) | 173 (173) | 64 (64) | 244 (244) | 79 (79)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 14 (15) | 5 (5)
Pain (General disorders) | 203 (203) | 66 (66) | 248 (249) | 77 (77)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 6 (8)
Pyrexia (General disorders) | 138 (138) | 51 (51) | 215 (219) | 65 (65)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2) | 11 (11) | 5 (5)
Somnolence (Nervous system disorders) | 90 (90) | 32 (32) | 190 (190) | 66 (66)
Swelling (General disorders) | 92 (92) | 32 (32) | 158 (158) | 52 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.